CLINICAL TRIAL: NCT02006641
Title: Randomised, Double-blind, Parallel-group, Placebo-controlled, Fixed-dose Study of Idalopirdine in Patients With Mild-moderate Alzheimer's Disease Treated With Donepezil
Brief Title: Idalopirdine in Patients With Mild-moderate Alzheimer's Disease Treated With Donepezil
Acronym: STARBEAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14862A; 2012-004764-22 (EudraCT Number)
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Results first posted 2018-02-20 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — (2-(6-fluoro-1H-indol-3-yl)-ethyl)-(3-(2,2,3,3-tetrafluoropropoxy)benzyl)amine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo adjunct to 10 mg Donepezil
  Interventions: Drug: Placebo
- Idalopirdine 10 mg (Experimental): Idalopirdine adjunct to 10 mg Donepezil
  Interventions: Drug: Idalopirdine
- Idalopirdine 30 mg (Experimental): Idalopirdine adjunct to 10 mg Donepezil
  Interventions: Drug: Idalopirdine

INTERVENTIONS:
Drug: Placebo — Once daily, matching placebo capsules, orally
  Arms: Placebo
Drug: Idalopirdine — Once daily, encapsulated tablets, orally
  Other Names: Lu AE58054
  Arms: Idalopirdine 10 mg; Idalopirdine 30 mg

SUMMARY:
To establish efficacy of Idalopirdine as adjunctive therapy to donepezil for symptomatic treatment of patients with mild-to-moderate Alzheimer's disease (AD).

DETAILED DESCRIPTION:
The study consisted of a screening period (up to 2-week period from screening to randomization), a 24-week double-blind treatment period with placebo or idalopirdine 10 mg/day or 30 mg/day as adjunctive therapy to donepezil 10 mg/day, and a 4-week safety follow-up period following study completion or withdrawal from treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a knowledgeable and reliable caregiver.
* The patient is an outpatient.
* The patient has probable AD.
* The patient has mild to moderate AD.
* Stable treatment with donepezil.
* The patient, if a woman, must have had her last natural menstruation ≥24 months prior to baseline, OR be surgically sterile.
* The patient, if a man, agrees to protocol-defined use of effective contraception if his female partner is of childbearing potential, OR must have been surgically sterilised prior to the screening visit.

Exclusion Criteria:

* The patient has evidence of any clinically significant neurodegenerative disease, or other serious neurological disorders other than AD.
* The patient has a Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM-IV-TR) Axis I disorder other than AD.
* The patient has evidence of clinically significant disease.
* The patient's donepezil therapy is likely to be interrupted or discontinued during the study.
* The patient is currently receiving memantine or has taken memantine within 2 months prior to screening.

Other inclusion and exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 858 (Actual)
Dates: Start 2014-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (162):
- United States (48):
  - US338, Phoenix, Arizona
  - US342, Fayetteville, Arkansas
  - US322, Anaheim, California
  - US305, Carson, California
  - US346, Costa Mesa, California
  - US327, Fullerton, California
  - US315, Lomita, California
  - US351, Oceanside, California
  - US307, Redlands, California
  - US301, Santa Rosa, California
  - US337, New London, Connecticut
  - US332, Stamford, Connecticut
  - US308, Delray Beach, Florida
  - US320, Hallandale, Florida
  - US347, Hialeah, Florida
  - US340, Lake Worth, Florida
  - US303, Miami, Florida
  - US313, Miami, Florida
  - US335, Naples, Florida
  - US345, Orange City, Florida
  - US309, Palm Beach Gardens, Florida
  - US302, Sunrise, Florida
  - US304, Atlanta, Georgia
  - US360, Augusta, Georgia
  - US318, Decatur, Georgia
  - US334, Lake Charles, Louisiana
  - US350, Belmont, Massachusetts
  - US344, Boston, Massachusetts
  - US310, Saint Paul, Minnesota
  - US321, Hattiesburg, Mississippi
  - US330, Creve Coeur, Missouri
  - US339, Paterson, New Jersey
  - US312, Staten Island, New York
  - US316, Charlotte, North Carolina
  - US336, Winston-Salem, North Carolina
  - US323, Cincinnati, Ohio
  - US349, Cleveland, Ohio
  - US306, Columbus, Ohio
  - US352, Lakewood, Ohio
  - US333, Oklahoma City, Oklahoma
  - US314, Allentown, Pennsylvania
  - US324, Pittsburgh, Pennsylvania
  - US341, Pittsburgh, Pennsylvania
  - US325, Reading, Pennsylvania
  - US319, Port Royal, South Carolina
  - US356, Cordova, Tennessee
  - US343, Fort Worth, Texas
  - US354, Houston, Texas
- Argentina (15):
  - AR303, Banfield
  - AR312, Buenos Aires
  - AR301, Ciudad Autonoma Buenos Aires
  - AR304, Ciudad Autonoma Buenos Aires
  - AR308, Ciudad Autonoma Buenos Aires
  - AR311, Ciudad Autonoma Buenos Aires
  - AR313, Ciudad Autonoma Buenos Aires
  - AR314, Ciudad Autonoma Buenos Aires
  - AR315, Ciudad Autonoma Buenos Aires
  - AR307, Córdoba
  - AR309, Córdoba
  - AR305, Godoy Cruz
  - AR310, Mendoza
  - AR302, Santa Fe
  - AR306, Santiago del Estero
- Brazil (5):
  - BR307, Curitiba
  - BR309, Curitiba
  - BR301, Rio de Janeiro
  - BR306, Rio de Janeiro
  - BR308, São Paulo
- Canada (6):
  - CA301, Halifax
  - CA302, Kelowna
  - CA306, Montreal
  - CA304, Qubec
  - CA303, Sherbrooke
  - CA305, Toronto
- Croatia (4):
  - HR304, Zabok
  - HR301, Zagreb
  - HR302, Zagreb
  - HR303, Zagreb
- Czechia (10):
  - CZ305, Brno
  - CZ306, Choceň
  - CZ309, Choceň
  - CZ308, Pardubice
  - CZ301, Prague
  - CZ303, Prague
  - CZ304, Prague
  - CZ307, Prague
  - CZ310, Praha 10 - Strasnice
  - CZ302, Rychnov nad Kněžnou
- Estonia (3):
  - EE301, Tallinn
  - EE303, Tallinn
  - EE302, Tartu
- Finland (3):
  - FI302, Kuopio
  - FI303, Oulu
  - FI301, Turku
- France (9):
  - FR301, Bordeaux
  - FR308, Bron
  - FR307, Colmar
  - FR304, Dijon
  - FR309, Élancourt
  - FR302, Marseille
  - FR303, Nice
  - FR306, Reims
  - FR305, Rouen
- Hungary (5):
  - HU304, Budapest
  - HU305, Budapest
  - HU301, Esztergom
  - HU303, Győr
  - HU302, Szeged
- IE301, Cork, Ireland
- Israel (3):
  - IL302, Haifa
  - IL303, Holon
  - IL304, Ramat Gan
- Italy (12):
  - IT306, Brescia
  - IT309, Brescia
  - IT311, Genova
  - IT312, Monza
  - IT302, Naples
  - IT313, Palermo
  - IT307, Perugia
  - IT301, Pisa
  - IT305, Roma
  - IT308, Roma
  - IT304, Torino
  - IT310, Torrette
- Lithuania (4):
  - LT302, Kaunas
  - LT303, Kaunas
  - LT301, Vilnius
  - LT304, Vilnius
- Poland (9):
  - PL301, Bialystok
  - PL304, Bydgoszcz
  - PL308, Gdynia
  - PL309, Krakow
  - PL302, Lodz
  - PL310, Lubin
  - PL306, Lublin
  - PL307, Oświęcim
  - PL303, Poznan
- Portugal (2):
  - PT301, Amadora
  - PT302, Coimbra
- South Korea (9):
  - KR303, Busan
  - KR301, Incheon
  - KR308, Seongnam-si
  - KR302, Seoul
  - KR304, Seoul
  - KR305, Seoul
  - KR306, Seoul
  - KR307, Seoul
  - KR309, Seoul
- Taiwan (5):
  - TW301, Kaohsiung City
  - TW302, Kaohsiung City
  - TW303, Taichung
  - TW304, Taipei
  - TW305, Taipei
- United Kingdom (9):
  - GB307, Amersham
  - GB301, Glasgow
  - GB303, London
  - GB308, London
  - GB306, Plymouth
  - GB305, Preston
  - GB304, Southampton
  - GB302, Swindon
  - GB309, Warrington

REFERENCES:
- [Derived] Ballard C, Atri A, Boneva N, Cummings JL, Frolich L, Molinuevo JL, Tariot PN, Raket LL. Enrichment factors for clinical trials in mild-to-moderate Alzheimer's disease. Alzheimers Dement (N Y). 2019 May 20;5:164-174. doi: 10.1016/j.trci.2019.04.001. eCollection 2019. PMID 31193334
- [Derived] Cummings JL, Atri A, Ballard C, Boneva N, Frolich L, Molinuevo JL, Raket LL, Tariot PN. Insights into globalization: comparison of patient characteristics and disease progression among geographic regions in a multinational Alzheimer's disease clinical program. Alzheimers Res Ther. 2018 Nov 24;10(1):116. doi: 10.1186/s13195-018-0443-2. PMID 30474567
- [Derived] Atri A, Frolich L, Ballard C, Tariot PN, Molinuevo JL, Boneva N, Windfeld K, Raket LL, Cummings JL. Effect of Idalopirdine as Adjunct to Cholinesterase Inhibitors on Change in Cognition in Patients With Alzheimer Disease: Three Randomized Clinical Trials. JAMA. 2018 Jan 9;319(2):130-142. doi: 10.1001/jama.2017.20373. PMID 29318278

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Idalopirdine 10 mg | Idalopirdine 30 mg
Started | 284 | 290 | 284
Treated | 282 | 285 | 281
Completed | 258 | 257 | 248
Not Completed | 26 | 33 | 36
Not completed — Withdrawal before treatment | 2 | 5 | 3
Not completed — Adverse Event | 15 | 11 | 15
Not completed — Protocol Violation | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 12 | 11
Not completed — Other reason: patient didn't show up | 1 | 0 | 0
Not completed — Other reason:patient didn't want to come | 0 | 0 | 1
Not completed — Other reason: patient has moved | 1 | 0 | 1
Not completed — Other reason: caregiver in hospital | 0 | 1 | 0
Not completed — Other reason: patient's wife has died | 0 | 0 | 1
Not completed — Other reason: hospitalisation | 0 | 1 | 0
Not completed — Other reason: caregiver impossibility | 0 | 0 | 1
Not completed — Other reason: protocol non-compliance | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: A total of 858 patients were randomized into the study but 10 patients were not treated (did not receive IMP). The baseline analysis population only consist of patients who have been treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Idalopirdine 10 mg | Idalopirdine 30 mg | Total
Number analyzed (Participants) | 282 | 285 | 281 | 848
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.4 (8.3) | 74.9 (8.1) | 75.0 (8.0) | 74.4 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181 | 172 | 169 | 522
  Male | 101 | 113 | 112 | 326
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 11 | 10 | 31
  Not Hispanic or Latino | 42 | 47 | 41 | 130
  Unknown or Not Reported | 230 | 227 | 230 | 687
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | NA — Information has not been collected | NA — Information has not been collected | NA — Information has not been collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian | 20 | 24 | 24 | 68
  Native Hawaiian or Other Pacific Islander | NA — Information has not been collected | NA — Information has not been collected | NA — Information has not been collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American | 6 | 6 | 4 | 16
  White | 250 | 249 | 244 | 743
  More than one race | NA — Information has not been collected | NA — Information has not been collected | NA — Information has not been collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 6 | 6 | 9 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 23 | 26 | 24 | 73
  Hungary | 7 | 4 | 4 | 15
  Czechia | 16 | 15 | 17 | 48
  United States | 54 | 58 | 52 | 164
  United Kingdom | 29 | 28 | 25 | 82
  Portugal | 4 | 6 | 5 | 15
  Canada | 11 | 9 | 10 | 30
  South Korea | 14 | 16 | 16 | 46
  Finland | 4 | 5 | 4 | 13
  Taiwan | 6 | 5 | 6 | 17
  Brazil | 13 | 13 | 11 | 37
  Poland | 31 | 26 | 30 | 87
  Italy | 21 | 22 | 22 | 65
  Israel | 3 | 3 | 3 | 9
  France | 12 | 12 | 12 | 36
  Lithuania | 13 | 16 | 16 | 45
  Estonia | 15 | 17 | 18 | 50
  Croatia | 6 | 4 | 6 | 16
MMSE total score at screening [Mean (Standard Deviation); unit: units on a scale] — The Mini Mental State Examination (MMSE) is an 11-item test to assess the cognitive aspects of mental function. The subtests assess orientation, memory, attention, language, and visual construction. The scores for each item is dichotomous (1 = response is correct, 0 = response is incorrect). Total score of the 11 items ranges from 0 to 30 (higher score indicates lower deficit).
  units on a scale | 17.6 (2.9) | 17.4 (3.0) | 17.5 (3.0) | 17.5 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognition
Description: Change from baseline to Week 24 in Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog) total score.
  The Alzheimer's Disease Assessment Scale - Cognitive subscale (ADAS-cog) is a 11-item neuropsychological test that assess the severity of cognitive impairment. The items determine the patient's orientation, memory, language, and praxis. Total score of the 11 items range from 0 to 70 (lower score indicates lower cognitive impairment).
Time Frame: Baseline and Week 24
Population: All patients who took at least one dose of placebo or idalopirdine, and who had a valid baseline assessment and at least one valid post-baseline assessment of the primary outcome measure in the 24-week treatment period (Full-analysis Set). For secondary outcome measures, the number of participants who had the respective outcome measure assessed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Idalopirdine 10 mg | Idalopirdine 30 mg
Number analyzed (Participants) | 278 | 282 | 275
units on a scale | 0.64 (0.39) | 0.55 (0.39) | 1.27 (0.39)
Statistical Analysis 1: Comparison: Placebo vs Idalopirdine 10 mg; For demonstrating efficacy of a dose, change in cognition (ADAS-cog) and either change in daily functioning (ADCS-ADL23) or change in global clinical impression (ADCS-CGIC) at Week 24 had to show statistically significant favourable differences compared to placebo at Week 24. Overall, type 1 error was controlled at 5% by multiplicity adjustment. Testing of the doses was done in a gated manner, first testing 30 mg at a 5% significance level, and only if found efficacious, then moving on to 10 mg; Test type: Superiority; p = 1.000, Mixed Models Analysis — Corrected for multiplicity; Treatment, country, MMSE stratum, week as fixed effects, baseline score, treatment-by-week, MMSE stratum-by-week, and baseline-by-week interactions; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-1.10 to 0.92], Standard Error of Mean 0.51 — A negative mean difference indicates a treatment effect in favour of idalopirdine
Statistical Analysis 2: Comparison: Placebo vs Idalopirdine 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.2223, Mixed Models Analysis — Corrected for multiplicity according to the multiple testing procedure; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.63, 95% CI 2-sided [-0.38 to 1.65], Standard Error of Mean 0.52 — A negative mean difference indicates a treatment effect in favour of idalopirdine

2. Secondary Outcome: Change in Daily Functioning
Description: Change from baseline to Week 24 in Alzheimer's Disease Cooperative Study - Activities of Daily Living Inventory (ADCS-ADL23) total score.
  The Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL23) is a 23-item clinician-rated inventory to assess activities of daily living (conducted with a caregiver or informant). Each item comprises a series of hierarchical sub-questions, ranging from the highest level of independent performance to a complete loss for each activity. Total score of the 23 items ranges from 0 to 78 (higher score indicates lower disability).
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Idalopirdine 10 mg | Idalopirdine 30 mg
Number analyzed (Participants) | 278 | 282 | 275
units on a scale | -1.39 (0.49) | -1.22 (0.49) | -1.36 (0.49)
Statistical Analysis 1: Comparison: Placebo vs Idalopirdine 10 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 1.000, Mixed Models Analysis — Corrected for multiplicity according to the multiple testing procedure; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.17, 95% CI 2-sided [-1.11 to 1.46], Standard Error of Mean 0.65 — A positive mean difference indicates a treatment effect in favour of idalopirdine
Statistical Analysis 2: Comparison: Placebo vs Idalopirdine 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 1.000, Mixed Models Analysis — Corrected for multiplicity according to the multiple testing procedure; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-1.27 to 1.33], Standard Error of Mean 0.66 — A positive mean difference indicates a treatment effect in favour of idalopirdine

3. Secondary Outcome: Change in Global Impression
Description: Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS-CGIC) score at Week 24.
  The Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change is a semi-structured interview to assess clinically relevant changes in patients with AD. The items determine cognition, behavior, social and daily functioning. Severity at baseline is rated on a 7-point scale from 1 (normal, not ill at all) to 7 (among the most extremely ill patients). The clinically relevant change from baseline is rated on a 7-point scale from 1 (marked improvement) to 7 (marked worsening).
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Idalopirdine 10 mg | Idalopirdine 30 mg
Number analyzed (Participants) | 277 | 282 | 275
units on a scale | 4.30 (0.06) | 4.24 (0.06) | 4.35 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Idalopirdine 10 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 1.000, Mixed Models Analysis — Corrected for multiplicity according to the multiple testing procedure; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.23 to 0.10], Standard Error of Mean 0.08 — A negative mean difference indicates a treatment effect in favour of idalopirdine
Statistical Analysis 2: Comparison: Placebo vs Idalopirdine 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 1.000, Mixed Models Analysis — Corrected for multiplicity according to the multiple testing procedure; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.12 to 0.21], Standard Error of Mean 0.09 — A negative mean difference indicates a treatment effect in favour of idalopirdine

4. Secondary Outcome: Change in Behavioural Disturbance
Description: Change from baseline to Week 24 in Neuropsychiatric Inventory (NPI) total score.
  The Neuropsychiatric Inventory is a 12-item structured interview with a caregiver to assess behavioural disturbances. The NPI comprises 10 behavioural and 2 neurovegetative items. Each item consists of a screening question and several sub-questions that are rated no (not present) or yes (present). Each item is rated for frequency (a 4-point scale from 1 [occasionally] to 4 [very frequent]) and severity (a 3-point scale from 1 [mild] to 3 [marked]). The total NPI score is the frequency ratings multiplied by the severity ratings and ranges from 0 to 144 (higher score indicates worse outcome).
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Idalopirdine 10 mg | Idalopirdine 30 mg
Number analyzed (Participants) | 278 | 282 | 275
units on a scale | -0.31 (0.59) | -0.94 (0.59) | -0.54 (0.60)

5. Secondary Outcome: Change in Individual Behavioural Disturbance Items
Description: Change in single NPI item scores at Week 24.
  The Neuropsychiatric Inventory is a 12-item structured interview with a caregiver to assess behavioural disturbances. The NPI comprises 10 behavioural and 2 neurovegetative items. Each item consists of a screening question and several sub-questions that are rated no (not present) or yes (present). Each item is then rated for frequency (a 4-point scale from 1 [occasionally] to 4 [very frequent]) and severity (a 3-point scale from 1 [mild] to 3 [marked]). Total score for each single NPI item ranges from 0-12 (frequency multiplied by severity), where higher scores represent worse outcome.
Time Frame: Baseline and Week 24
Population: All patients who took at least one dose of placebo or idalopirdine and who had a valid baseline assessment and at least one valid post-baseline assessment of the primary outcome measure in the 24-week treatment period (Full-analysis Set). For secondary outcome measures, the number of participants who had the respective outcome measure/item assessed
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Idalopirdine 10 mg | Idalopirdine 30 mg
Number analyzed (Participants) | 278 | 282 | 275
units on a scale
  Delusions | 0.01 (0.08) | -0.18 (0.08) | 0.00 (0.08)
  Hallucinations | 0.00 (0.04) | -0.06 (0.04) | -0.03 (0.04)
  Agitation/aggression | 0.02 (0.11) | -0.06 (0.11) | -0.06 (0.11)
  Depression/dysphoria | -0.20 (0.10) | -0.08 (0.10) | -0.14 (0.10)
  Anxiety | -0.05 (0.11) | -0.06 (0.11) | -0.02 (0.11)
  Elation/euphoria | 0.01 (0.04) | -0.05 (0.04) | -0.02 (0.04)
  Apathy/indifference | 0.00 (0.17) | -0.19 (0.17) | -0.24 (0.17)
  Disinhibition | 0.08 (0.09) | -0.04 (0.09) | 0.02 (0.09)
  Irritability/lability | 0.03 (0.12) | -0.05 (0.12) | -0.17 (0.12)
  Aberrant motor behaviour | -0.03 (0.14) | 0.06 (0.14) | 0.12 (0.14)
  Sleep | -0.04 (0.12) | -0.07 (0.12) | 0.12 (0.12)
  Appetite/eating disorder | -0.14 (0.14) | -0.30 (0.14) | -0.07 (0.14)

6. Secondary Outcome: Change in NPI Anxiety Item Score in Patients With an NPI Anxiety Item Score of at Least 2 at Baseline
Description: Change from baseline to Week 24 in NPI anxiety item score in patients with an NPI anxiety item score of at least 2 at baseline
  The Neuropsychiatric Inventory is a 12-item structured interview with a caregiver to assess behavioural disturbances. The NPI comprises 10 behavioural and 2 neurovegetative items. Each item consists of a screening question and several sub-questions that are rated no (not present) or yes (present). Each item is then rated for frequency (a 4-point scale from 1 [occasionally] to 4 [very frequent]) and severity (a 3-point scale from 1 [mild] to 3 [marked]). The total score for the NPI anxiety item ranges from 0-12 (frequency multiplied by severity), where a higher score represents a worse outcome.
Time Frame: Baseline and Week 24
Population: All patients who took at least one dose of placebo or idalopirdine and who had a valid baseline assessment and at least one valid post-baseline assessment of the primary outcome measure in the 24-week treatment period (Full-analysis Set). For secondary outcome measures, the number of participants who had the respective outcome/item measure assessed
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Idalopirdine 10 mg | Idalopirdine 30 mg
Number analyzed (Participants) | 71 | 56 | 61
units on a scale | -1.48 (0.38) | -1.82 (0.40) | -1.69 (0.40)

7. Secondary Outcome: Number of Participants With Clinical Improvement
Description: Clinical response at Week 24 (based on pre-specified ADAS-cog, ADCS-ADL23, and ADCS-CGIC changes [change in ADAS-cog below or equal to -4, change in ADCS-ADL23 at least 0, and ADCS-CGIC below or equal to 4])
Time Frame: Week 24
Population: All patients who took at least one dose of placebo or idalopirdine and who had a valid baseline assessment and at least one valid post-baseline assessment of the primary outcome measure in the 24-week treatment period (Full-analysis Set). For secondary outcome measures, the number of participants who had the respective outcome measure assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Idalopirdine 10 mg | Idalopirdine 30 mg
Number analyzed (Participants) | 255 | 257 | 249
Participants | 20 | 33 | 22

8. Secondary Outcome: Number of Participants With Clinical Worsening
Description: Clinical worsening at Week 24 (Based on pre-specified ADAS-cog, ADCS-ADL23, and ADCS-CGIC changes [change in ADAS-cog above or equal to 4, change in ADCS-ADL23 below 0, and ADCS-CGIC above 4])
Time Frame: Week 24
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Idalopirdine 10 mg | Idalopirdine 30 mg
Number analyzed (Participants) | 255 | 257 | 249
Participants | 27 | 28 | 27

9. Secondary Outcome: Change in Cognitive Aspects of Mental Function
Description: Change from baseline to Week 24 in Mini Mental State Examination (MMSE). The Mini Mental State Examination (MMSE) is an 11-item test to assess the cognitive aspects of mental function. The subtests assess orientation, memory, attention, language, and visual construction. The scores for each item is dichotomous (1 = response is correct, 0 = response is incorrect). Total score of the 11 items ranges from 0 to 30 (higher score indicates lower deficit).
Time Frame: Baseline and Week 24
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Idalopirdine 10 mg | Idalopirdine 30 mg
Number analyzed (Participants) | 258 | 257 | 248
units on a scale | -0.24 (0.21) | -0.45 (0.21) | -0.34 (0.21)

10. Secondary Outcome: Change in Health-related Quality of Life (EQ-5D) Utility Score
Description: Change from baseline to Week 24 in EuroQol 5-dimensional (EQ-5D) utility score
  The EQ-5D is a patient-reported assessment that measures the patient's well-being. It consists of an utility score based on 5 descriptive items (mobility, self-care, usual activities, pain/discomfort, and depression/anxiety) and a Visual Analogue Scale (VAS). Each descriptive item is rated on a 3-point index ranging from 1 (no problems) to 3 (extreme problems) that is used for calculating a single summary index (from 0 to 1). A higher EQ-5D score indicates a worse outcome.
Time Frame: Baseline and Week 24
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Idalopirdine 10 mg | Idalopirdine 30 mg
Number analyzed (Participants) | 274 | 275 | 266
units on a scale | 0.03 (0.01) | 0.02 (0.01) | 0.01 (0.01)

11. Secondary Outcome: Change in Health-related Quality of Life (EQ-5D VAS)
Description: Change from baseline to Week 24 in EQ-5D Visual Analogue Scale (EQ-5D VAS).
  The EQ-5D is a patient-reported assessment that measures the patient's well-being. It consists of an utility score based on 5 descriptive items (mobility, self-care, usual activities, pain/discomfort, and depression/anxiety) and a Visual Analogue Scale (VAS). The VAS ranges from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Baseline and Week 24
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Idalopirdine 10 mg | Idalopirdine 30 mg
Number analyzed (Participants) | 274 | 274 | 266
units on a scale | 1.35 (0.99) | 1.87 (0.99) | 1.00 (1.01)

ADVERSE EVENTS:
Time Frame: Baseline to end of study at Week 24
Description: Treatment-Emergent Adverse Events are reported in this section
Groups:
- Idalopirdine 30 mg: Idalopirdine adjunct to 20 mg Donepezil
  Idalopirdine: Once daily, encapsulated tablets, orally
Arm/Group | Placebo | Idalopirdine 10 mg | Idalopirdine 30 mg
All-Cause Mortality (participants affected / at risk) | 1/282 | 0/285 | 1/281
Serious Adverse Events (participants affected / at risk) | 12/282 | 13/285 | 15/281
Other Adverse Events (participants affected / at risk) | 33/282 | 26/285 | 31/281
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=282) | Idalopirdine 10 mg (N=285) | Idalopirdine 30 mg (N=281)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 2
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Carotid sinus syndrome (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 0
Dementia (Nervous system disorders) | 1 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 2 | 0 | 1
Depressive symptom (Psychiatric disorders) | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Hallucinations, mixed (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/101 | 0/113 | 1/112
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=282) | Idalopirdine 10 mg (N=285) | Idalopirdine 30 mg (N=281)
Accidental overdose (Injury, poisoning and procedural complications) | 33 | 26 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No